CLINICAL TRIAL: NCT06013267
Title: Effects of Chin Tuck Against Resistance Exercise on Patients With Dysphagia After Stroke: A Randomized Controlled Trial
Brief Title: Effects of Chin Tuck Against Resistance Exercise on Patients With Dysphagia After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chia-Chi Kuo, Associate Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUAN20230103B
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: stroke; dysphagia; chin tuck against resistance exercise; randomized controlled trial
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will receive a four-week "CTAR exercise protocol " and routine dysphagia care.
  Interventions: Other: Chin tuck against resistance exercise
- control group (No Intervention): The control group will only receive routine dysphagia care.

INTERVENTIONS:
Other: Chin tuck against resistance exercise — The experimental group will receive a four-week CTAR protocol and regular dysphagia care, while the control group will only receive routine dysphagia care. The routine dysphagia care is including dysphagia education, dietary precautions, oral hygiene, and swallowing training, etc. The CTAR protocol is first, the study nurses face-to-face teach dysphagia patients to perform CTAR exercises once, then the patient perform CTAR exercises three times a day, five days a week, and for four weeks. The CTAR exercise is to tighten a rubber ball which placed between the chin and the sternum, and to perform 3 cycles of isometric exercise and isotonic exercise.
  Other Names: Routine dysphagia care
  Arms: experimental group

SUMMARY:
The aim of this clinical trial is to explore the effects of chin tuck against resistance (CTAR) exercises on improving dysphagia in stroke patients.

The main aims of this research are:

1. To explore the effects of CTAR exercise on stroke patients with dysphagia, and to perform a clinically implementable evidence-based protocol.
2. Introduce the evidence-based "CTAR exercise protocol" in the care of stroke patients with dysphagia, and test the effects through a randomized controlled trial.

This study is a two-group, pre and post-test, parallel, non-blind randomized controlled trial to test the effectiveness of the "CTAR exercise protocol". Convenience sampling the inpatients of stroke with dysphagia from a regional hospital in southern Taiwan. Eighty participants will be randomized block assignment either to an experimental (n = 40) or to a control (n = 40) group. The experimental group will receive a four-week CTAR protocol and regular dysphagia care. The control group will receive the regular dysphagia care only. In this study, dysphagia-related physiological indicators including functional oral intake scale (FOIS), penetration-aspiration scale (PAS), and modified water swallowing test, video fluoroscopic swallowing study (VFSS), and swallowing improvement rate will be used to evaluate the difference between pre-test and four-week post-test after the intervention. The independent t-test will be used to compare the change effect of the two groups.

DETAILED DESCRIPTION:
This study is a two-group, pre- and post-test, parallel, non-blind randomized controlled trial to test the effectiveness of the "chin retraction resistance exercise program". The convenient sampling will be used to select inpatients with stroke and dysphagia in a regional hospital from southern Taiwan. In this study, the investigators will use block randomization to assign participants to either experimental or control group, and use sealed opaque envelopes to conceal the allocation sequences. The target sample size of 80 participants will be enrolled according to sample size calculation. The CTAR exercise is to tighten a rubber ball which placed between the chin and the sternum, and to perform 3 cycles of isometric exercise and isotonic exercise. The CTAR protocol is perform CTAR exercises three times a day, five days a week, and for four weeks. The research nurses will assist in screen and recruit subjects in clinical ward units, perform the CTAR exercise protocol, and collect dates. The independent t-test will be used to compare the change effect of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with newly diagnosed stroke with dysphagia.
* The modified water swallowing test shows that ≦ 4 points, which mean patient have a high risk of swallowing disorders.
* Adults over 20 years old, without visual, hearing and mental disabilities.
* Patients who have clear consciousness and can sit up at least 10 minutes to cooperate with swallowing training.

Exclusion Criteria:

* In addition to not meeting the above selection criteria, those who have head and neck cancer or movement disorders and cannot cooperate with the chin tuck against resistance exercise will be listed as excluded cases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The functional oral intake scale: One question, 1~7 scores. | Pre-test and four-week post-test
  The functional oral intake scale (FOIS) is a 7-point scale, which is used to measure the state of eating by mouth. A score of 1 means that patient can't eat by mouth at all, and a score of 7 means patient can eat food of any stickiness and type by mouth. The research nurse will use this scale to test the state of eating by mouth of participants, and collect the pre-test and four-week post-test data then record on an excel dataset.
The penetration-aspiration scale: One question, 1~8 scores. | Pre-test and four-week post-test
  The penetration-aspiration scale (PAS) is an 8-point scale used to measure laryngeal leakage and aspiration severity, which with higher scores representing more severe respiratory aspiration. A score of 1 means that normal swallowing function, and a score of 8 means food mistakenly enters airway and without cough re¬flex during swallowing. The research nurse will use this scale to test the laryngeal leakage and aspiration severity of participants, and collect the pre-test and four-week post-test data then record on an excel dataset.
The modified water swallowing test : One question, 1~5 scores. | Pre-test and four-week post-test
  The modified water swallowing test (MWST) is a 1 to 5-point scale, which is a routine used clinical swallowing test. The researcher nurse will inject 3ml of cold water into the bottom of the participant's mouth with an injection syringe, and then asks the participant to swallow the water for the swallowing test. If the participant is unable to swallow, or experienced dyspnea, coughing, or wet-hoarse dysphonia after swallowing, a score of 1-3 will be respective recorded. The lower the score, meaning the more serious problem of swallowing and choking. The sensitivity and specificity of MWST to differentiate between aspirators and non-aspirators with a cutoff level of 3 are 70 and 88%, respectively. The research nurse will use this scale to test the water swallowing function of participants for a screen scale of inclusion criteria, and collect the pre-test and four-week post-test data then record on an excel dataset.
video fluoroscopic swallowing study (VFSS) | Pre-test and four-week post-test
  The video fluoroscopic swallowing study (VFSS) is a routine clinical swallowing photography examination to diagnosis the dysphagia problems and severity, which is perform and report by radiologist. The radiologist will interpret the image and report the swallowing function of VFSS as normal, penetration, or aspiration. The research nurse will collect the data of swallowing function on the existing VFSS reports of the electronic medical records. The collected measurement data will be aggregated on an excel dataset.photography examination, and the research nurse will collect the existing VFSS report on the electronic medical records.

SECONDARY OUTCOMES:
The swallowing improvement rate: Number of participants with swallowing improvement event as assessed by the modified water swallowing test. | Four-week post-test
  Based on the pre- and post-test scores of the modified water drinking test, the researcher will calculate the number of participants who have present improved at post-test scores, and then calculate the swallowing improvement rates of the two groups. The formula is: The swallowing improvement rate= Number of participants with improve events (modified water swallowing test showed the post-test score is improve compare to pre-test) ÷ number of participants of each group × 100%.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao J, Zhang HJ. Effects of chin tuck against resistance exercise versus Shaker exercise on dysphagia and psychological state after cerebral infarction. Eur J Phys Rehabil Med. 2017 Jun;53(3):426-432. doi: 10.23736/S1973-9087.16.04346-X. Epub 2016 Nov 10. PMID 27830923
- [Background] Kim HH, Park JS. Efficacy of modified chin tuck against resistance exercise using hand-free device for dysphagia in stroke survivors: A randomised controlled trial. J Oral Rehabil. 2019 Nov;46(11):1042-1046. doi: 10.1111/joor.12837. Epub 2019 Jul 2. PMID 31206210
- [Background] Oguchi N, Yamamoto S, Terashima S, Arai R, Sato M, Ikegami S, Horiuchi H. The modified water swallowing test score is the best predictor of postoperative pneumonia following extubation in cardiovascular surgery: A retrospective cohort study. Medicine (Baltimore). 2021 Jan 29;100(4):e24478. doi: 10.1097/MD.0000000000024478. PMID 33530263
- [Background] Dziewas R, Michou E, Trapl-Grundschober M, Lal A, Arsava EM, Bath PM, Clave P, Glahn J, Hamdy S, Pownall S, Schindler A, Walshe M, Wirth R, Wright D, Verin E. European Stroke Organisation and European Society for Swallowing Disorders guideline for the diagnosis and treatment of post-stroke dysphagia. Eur Stroke J. 2021 Sep;6(3):LXXXIX-CXV. doi: 10.1177/23969873211039721. Epub 2021 Oct 13. PMID 34746431
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Park JS, An DH, Oh DH, Chang MY. Effect of chin tuck against resistance exercise on patients with dysphagia following stroke: A randomized pilot study. NeuroRehabilitation. 2018;42(2):191-197. doi: 10.3233/NRE-172250. PMID 29562558
- [Background] Park JS, Lee G, Jung YJ. Effects of game-based chin tuck against resistance exercise vs head-lift exercise in patients with dysphagia after stroke: An assessor-blind, randomized controlled trial. J Rehabil Med. 2019 Oct 29;51(10):749-754. doi: 10.2340/16501977-2603. PMID 31515567
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037